CLINICAL TRIAL: NCT04131894
Title: Healing of Extraction Sockets Preserved With Autogenous Dentin Graft: A Clinical, Histological, Histomorphometrical and Electron Microscobic Study
Brief Title: Effects of Autogenous Dentin Graft on Socket Preservation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Collaborators: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Ezgi Yüceer Çetiner, Assistant Professor, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 71146310 [2015-AC-CE-42]
Record Dates: First submitted 2019-10-15; First posted 2019-10-18 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Bone Regeneration; Bone And Bones; Bone Substitutes
Keywords: augmentation; dentin graft; socket preservation

ARMS (3):
- Control (No Intervention): Extraction sockets with spontaneous healing (16 sockets).
- Dentin (Active Comparator): Extraction sockets were filled with undemineralized autogenous dentin graft (20 sockets).
  Interventions: Biological: autogenous dentin graft
- Dentin+PRF (Active Comparator): Extraction sockets were filled with mixture of undemineralized autogenous dentin graft and platelet rich fibrin (PRF) (21 sockets).
  Interventions: Biological: autogenous dentin graft; Biological: platelet rich fibrin (PRF)

INTERVENTIONS:
Biological: autogenous dentin graft
  Arms: Dentin; Dentin+PRF
Biological: platelet rich fibrin (PRF)
  Arms: Dentin+PRF

SUMMARY:
Various graft materials are used to reconstruct bone defects in the jaws due to tooth loss, trauma, advanced periodontal diseases, pathological lesions and congenital disorders. The main features of an ideal bone graft are osteogenesis, osteoinduction and osteoconduction. Autogenous bone graft is considered as the gold standard among all bone graft materials. Because it has all the features that an ideal bone graft should have. However, there are some disadvantages such as donor site morbidity, obtaining limited amounts and high rates of resorption. Because of these disadvantages, other bone graft materials such as allografts, xenografts and alloplastic bone grafts are frequently used for bone augmentation. In the light of recent studies, the limits of conventional bone graft materials such as limited osteoconduction capacity and disease transmission have been clearly demonstrated. Due to the disadvantages of these materials, studies are directed to develop alternative graft materials. Aim of this study is to analyse the effects of autogenous dentin graft and mixture of autogenous dentin graft and platelet rich fibrin (PRF) applied to the tooth extraction sockets on bone healing process. A total of 57 extraction sockets in 9 patients who were planned to be treated with dental implant after tooth extraction were evaluated in this study. Extraction sockets were divided randomly into 3 groups. In the first group, sockets were filled with autogenous dentin graft (Group D-20 sockets). In the second group, sockets were filled with the mixture of PRF and autogenous dentin graft (Group DP-21 sockets). In the third group, sockets were left empty as control group (Group C-16 sockets). After 3 months, histological and immunohistochemical evaluations were performed on the samples taken during the implant surgery. Additionally, samples obtained from each group were examined by scanning electron microscopy (SEM).

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years,
* Systemically healthy patients (ASA I and II),
* Adequate restorative space for implant-retained restoration.

Exclusion Criteria:

* Teeth with deep decay or root canal filling,
* Systemically complicated patients (ASA III, IV, V),
* Presence of acute infection,
* Pregnancy or lactation,
* Unwillingness to return for the follow-up periods

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-08-27 (Actual)

PRIMARY OUTCOMES:
Histopathological Evaluation | 3 months after the augmentation procedure
  Samples obtained from the groups were fixed in 10% formalin solution and decalcified in 5% formic acid solution. The samples were gradually dehydrated in an ethanol series, placed in xylene for clearing, and then embedded in paraffin. The tissue blocks were sectioned at 5µm on a rotary microtome (Leica RM 2125RT, Nussloch, Germany). Sections were stored overnight at 60°C for deparaffinization. Then the deparaffinization process was completed with xylene series. Following this procedure, the sections were passed from the alcohol series and dehydrated. Following deparaffinization, all sections were stained using Hematoxylin-Eosin staining method. Five sections were taken from each sample and used for histopathological evaluation. Images were taken from all sections in X4, X10 and X20 magnification using light microscope (Olympus BX43, Center Valley, PA) with camera attachment. New bone, connective tissue, graft and blood vessel volumes were evaluated by histopathological scoring method.
Immunohistochemical Evaluation | 3 months after the augmentation procedure
  Sections (5 µm) were taken from each sample and deparafinization was completed. Mouse and Rabbit Specific HRP / AEC (ABC) Detection IHC Kit (Abcam, USA) was used to perform the reactions. After this process, the sections were exposed until color change in order to show the immune reaction in the tissue and counterstained briefly with Mayer's hematoxylin. Anti-BMP-2 and anti-RUNX-2 antibodies (Abcam, USA) were used. Finally, the sections were washed with distilled water and then covered with immune closure medium. Images were taken in X4, X10, X20 magnification using light microscope (Olympus BX43, Center Valley, PA) with camera attachment (Carl Zeiss, Germany).
Scanning Electron Microscopy (SEM) Evaluation | 3 months after the augmentation procedure
  After the drying process, 4 samples from each group were coated with a 10 nm thick gold-palladium layer using the coating device (Balzers-SCd 050, Germany). The samples were analyzed at 10 kV with the SEM device (JSM-7001 F, JEOL, Tokyo, Japan) for the purpose of examining the surface formation. For each group, the image was taken at X2000, X5000 and X10.000 magnification.